CLINICAL TRIAL: NCT02872896
Title: The Role of Noninvasive Beat-to-Beat ClearSight Blood Pressure Monitoring During Non-cardiac Surgery
Brief Title: Noninvasive Beat-to-Beat ClearSight Blood Pressure Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Kamal Maheshwari, MD MPH, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16-845
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — Orthopedic Procedures; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ClearSight device (Experimental): Patients having orthopedic, urologic or general surgery will have blood pressure monitored by the ClearSight device second by second throughout surgery.
  Interventions: Procedure: Orthopedic, urologic or general surgery
- Non-ClearSight (Sham Comparator): Patients having orthopedic, urologic or general surgery will have blood pressure monitored by the Non-ClearSight (the clinical team) every 5 minutes throughout surgery.
  Interventions: Procedure: Orthopedic, urologic or general surgery

INTERVENTIONS:
Procedure: Orthopedic, urologic or general surgery — Patients having orthopedic, urologic or general surgery may have the ClearSight device; patients having orthopedic, urologic or general surgery may have the non-ClearSight device to monitor subject blood pressure during surgery

SUMMARY:
Subjects will first have a blood pressure reading recorded on both arms using a non-invasive blood pressure monitoring (NIBP) cuff in the preoperative area. Then blood pressure will be recorded using the ClearSight monitor on each hand over a one-minute period. If mean arterial pressure (MAP) as assessed by either the noninvasive blood pressure (NIBP) monitoring cuff or the ClearSight system differs by more than 10% from arm to arm, the subject will be excluded from the study.

Before induction of anesthesia, the subject will be randomized to either:

ClearSight group + usual clinical care: Information from ClearSight monitor will be available to the clinicians. According to ASA guidelines, usual blood pressure monitoring includes non-invasive blood pressure measurements every 5 minutes during a surgical case.

Non-ClearSight group (blinded) + usual clinical care: Information from ClearSight monitor will not be available to the clinicians.

Both patient groups will have continuous ClearSight monitoring and non-invasive blood pressure monitoring every 5 minutes. The difference will be in the intervention group data from the monitor will be available to the clinicians in the operating room, but in the control group data from the ClearSight monitor will not be available (blinded) to the clinicians. Regardless of the study group assignment, second-by-second ClearSight monitor continuous blood pressure data will be recorded for each study patient and will be used for analysis.

The morning of post-operative day 3 the subject will be given the QoR-15 questionnaire and will complete POMS morbidity surveys.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age > 45 years
* ASA Physical Status 3 or 4
* Moderate- or high-risk non-cardiac surgical procedures (i.e., orthopedic, spine, urology, and general surgery) in patients in whom invasive blood pressure monitoring is not planned
* Anticipated surgical duration >2 hours

Exclusion Criteria:

* Any contraindications to the proposed interventions
* Patient with invasive blood pressure monitoring
* Patients with contraindications to oscillometric blood pressure monitoring on one arm and ClearSite monitoring on the other
* Preoperative discrepancy in mean arterial pressure >10% between the arms

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2016-10; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Time- weighted average (TWA) MAP | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sessler, M.D., Study Chair — Department Chair
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Maheshwari K, Buddi S, Jian Z, Settels J, Shimada T, Cohen B, Sessler DI, Hatib F. Performance of the Hypotension Prediction Index with non-invasive arterial pressure waveforms in non-cardiac surgical patients. J Clin Monit Comput. 2021 Feb;35(1):71-78. doi: 10.1007/s10877-020-00463-5. Epub 2020 Jan 27. PMID 31989416
- [Derived] Maheshwari K, Khanna S, Bajracharya GR, Makarova N, Riter Q, Raza S, Cywinski JB, Argalious M, Kurz A, Sessler DI. A Randomized Trial of Continuous Noninvasive Blood Pressure Monitoring During Noncardiac Surgery. Anesth Analg. 2018 Aug;127(2):424-431. doi: 10.1213/ANE.0000000000003482. PMID 29916861